CLINICAL TRIAL: NCT00450411
Title: A Prospective Phase II Trial of Transperineal Ultrasound-Guided Brachytherapy for Locally Recurrent Prostate Adenocarcinoma Following External Beam Radiotherapy
Brief Title: Ultrasound-Guided Implant Radiation Therapy in Treating Patients With Locally Recurrent Prostate Cancer Previously Treated With External-Beam Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0526; CDR0000533887
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Iodine-125; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brachytherapy (Experimental): Prostate brachytherapy delivered using either 125-iodine (I-125) or 103-palladium (Pd-103)
  Interventions: Radiation: 125-Iodine; Radiation: 103-palladium

INTERVENTIONS:
Radiation: 125-Iodine — Brachytherapy to the prostate via 125-iodine (I-125) seeds with a planned dose of 140 Gy
  Other Names: brachytherapy
Radiation: 103-palladium — Brachytherapy to the prostate via 103-palladium (Pd-103) seeds with a planned dose of 120 Gy
  Other Names: brachytherapy

SUMMARY:
RATIONALE: Implant radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well ultrasound-guided implant radiation therapy works in treating patients with locally recurrent prostate cancer previously treated with external-beam radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the late treatment-related gastrointestinal (GI) and genitourinary (GU) adverse events in patients with locally recurrent adenocarcinoma of the prostate previously treated with external-beam radiotherapy who are currently receiving transperineal ultrasound-guided iodine I 125 or palladium Pd 103 brachytherapy.

Secondary

* Determine the acute treatment-related GI and GU adverse events in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the disease-free survival of patients treated with this regimen.
* Determine the disease-specific survival of patients treated with this regimen.
* Determine clinical patterns of tumor recurrence (time to local tumor progression or distant failure) in patients treated with this regimen.
* Determine the time to biochemical failure in patients treated with this regimen.
* Determine the post-brachytherapy dosimetric coverage in patients treated with this regimen.

OUTLINE: This is a prospective, multicenter study.

Patients undergo transperineal ultrasound-guided iodine I 125 or palladium Pd 103 brachytherapy.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 96 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-documented locally recurrent prostatic adenocarcinoma > 30 months after the completion of EBRT, biopsied ≤ 180 days prior to registration and confirmed by central pathology review
2. Disease-related characteristics at initial diagnosis (i.e., prior to EBRT) that fit the following criteria: Stages T1-T2c, Gleason scores 2-7, and PSA ≤ 20 ng/mL
3. Staging, performed within 8 weeks prior to registration:

   * 3.1 History/physical examination (to include at a minimum digital rectal examination of the prostate and examination of the skeletal system and abdomen)
   * 3.2 Negative lymph nodes by imaging (pelvic ± abdominal CT or MR), or by nodal dissection (laparoscopy or laparotomy)
   * 3.3 No evidence of bone metastases (M0) on bone scan
4. Zubrod Performance Scale 0-1
5. American Urological Association Symptom Index Score (AUA BPH) < 15 (Note: The use of alpha blockers is permitted when evaluating lower urinary tract symptoms, i.e., the AUA score with the patient on alpha blockers is acceptable)
6. Age ≥ 18
7. Baseline serum prostate-specific antigen (PSA) value < 10 ng/mL performed with an FDA-approved assay (e.g., Abbott, Hybritech) within 8 weeks prior to registration. PSA should not be performed within 10 days of a prior prostate biopsy, and if the patient has been started on hormonal therapy, the PSA should be performed within 8 weeks prior to the commencement of hormonal therapy.
8. Prostate volume as measured by transrectal ultrasound (TRUS) ≤ 45 cc or pubic arch interference ruled out
9. The patient must be suitable for spinal or general anesthesia
10. The patient must sign a study-specific informed consent form before study entry

Exclusion Criteria:

1. Prior invasive (except non-melanoma skin cancer) or hematological (e.g., acute leukemia, aggressive lymphoma, myeloma) malignancy unless disease-free for a minimum of 3 years. Previous diagnosis of low-grade lymphoma or chronic lymphocytic leukemia is allowed.
2. Prior EBRT to the prostate such that the minimum dose to the prostate exceeded 78 Gy (2 Gy fractions) or 79.8 Gy (1.9 Gy fractions) or 81 Gy (1.8 Gy fractions)
3. Baseline gastrointestinal (GI) or genitourinary (GU) toxicity (for any reason) grade ≥ 2 as defined in Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
4. Severe, active co-morbidity, defined as follows:

   * 4.1 Unstable angina and/or decompensated congestive heart failure
   * 4.2 Myocardial infarction within the last 6 months
   * 4.3 Bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * 4.4 Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   * 4.5 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   * 4.6 Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
5. Clinical and/or radiologic evidence of extraprostatic disease at initial diagnosis (i.e., prior to EBRT) or at time of local recurrence (i.e., prior to study registration)

   ° 5.1 Histologic or radiologic evidence of tumor involvement of regional lymph nodes (N1) or the presence of metastatic disease (M1)
6. Any of the following prior therapies:

   * Transurethral resection of the prostate (TURP)
   * Radionuclide (permanent or temporary implantation) prostate brachytherapy
   * Prostatectomy or prostatic cryosurgery
   * High-intensity focused ultrasound (HIFU)
   * Bilateral orchiectomy
   * Chemotherapy for prostatic carcinoma
   * NOTE 1: Androgen suppression therapy is permissible provided that the luteinizing hormone-releasing hormone (LHRH) agonist was started at least 2 months and no more than 6 months before registration.
   * NOTE 2: Any combination of neoadjuvant, concurrent, or adjuvant androgen suppression therapy at the time of initial external radiotherapy is permissible provided the total duration was ≤ 8 months. If > 8 months, evidence of a normal serum testosterone must be documented.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2016-06 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juanita M. Crook, MD, Study Chair — British Columbia Cancer Agency
Locations (17):
- United States (13):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - California Cancer Center - Woodward Park Office, Fresno, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Robinson Radiation Oncology, Ravenna, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
- Canada (4):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Crook J, Rodgers JP, Pisansky TM, Trabulsi EJ, Amin MB, Bice W, Morton G, Murtha AD, Vigneault E, Helou J, Michalski JM, Roach M 3rd, Beyer D, Jani AB, Horwitz EM, Raben A, Pugh S, Sandler H. Salvage Low-Dose-Rate Prostate Brachytherapy: Clinical Outcomes of a Phase 2 Trial for Local Recurrence after External Beam Radiation Therapy (NRG Oncology/RTOG 0526). Int J Radiat Oncol Biol Phys. 2022 Apr 1;112(5):1115-1122. doi: 10.1016/j.ijrobp.2021.10.138. Epub 2021 Nov 3. PMID 34740768
- [Derived] Crook JM, Zhang P, Pisansky TM, Trabulsi EJ, Amin MB, Bice W, Morton G, Pervez N, Vigneault E, Catton C, Michalski J, Roach M 3rd, Beyer D, Jani A, Horwitz E, Donavanik V, Sandler H. A Prospective Phase 2 Trial of Transperineal Ultrasound-Guided Brachytherapy for Locally Recurrent Prostate Cancer After External Beam Radiation Therapy (NRG Oncology/RTOG-0526). Int J Radiat Oncol Biol Phys. 2019 Feb 1;103(2):335-343. doi: 10.1016/j.ijrobp.2018.09.039. Epub 2018 Oct 9. PMID 30312717

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brachytherapy
Started | 100
Eligible and Started Protocol Treatment | 92
Completed (Subjects contributing data to analysis are considered to have completed the study.) | 92
Not Completed | 8
Not completed — Protocol Violation | 6
Not completed — No protocol treatment | 2

BASELINE CHARACTERISTICS:
Population: Eligible patients who received protocol treatment
Arm/Group | Brachytherapy
Number analyzed (Participants) | 92
Age, Continuous [Median (Full Range); unit: years] | 70 [55 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Late Treatment-related Gastrointestinal (GI) and Genitourinary (GU) Adverse Events (AE)
Description: Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. For the purposes of this study, late treatment-related adverse events were evaluated between 271 days and 730 days from the implant.
Time Frame: Between 271 days and 730 days from date of implantation
Population: Eligible patients who received protocol treatment with at least 23 months follow-up from the date of implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 87
Participants | 12
Statistical Analysis 1: Comparison: Brachytherapy; It was projected that ≤10% of patients would experience late treatment-related GI/GU AEs under the protocol treatment (alternative hypothesis). A rate of ≥20% was considered unacceptable (null hypothesis). With a one-sided significance level of 0.05, it was estimated that 87 analyzable patients were required to detect the above-mentioned effect size with an 85% statistical power using Fleming's multiple testing procedure with two interim analyses and one final analysis; Test type: Other; Stopping Rules for a Late GI/GU Adverse Event: For 44 patients, if ≤2 then reject H0, if ≥8 then reject HA; for 73 patients, if ≤7 then reject H0, if ≥10 then reject HA; for 87 patients, if ≤10 then reject H0, if ≥11 then reject HA

2. Secondary Outcome: Number of Patients With Acute Treatment-related GI and GU Adverse Events
Description: Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. For the purposes of this study, acute treatment-related adverse events will be evaluated within 270 days from the implant.
Time Frame: From date of implantation to 270 days
Population: Eligible patients who received protocol treatment with at least 270 days of follow-up from the date of implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 88
Participants | 12

3. Secondary Outcome: Percentage of Participants Alive at 5 Years (Overall Survival)
Description: Survival time is defined as time from registration to date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. Analysis occurred after all patients were potentially observed for at least 5 years from registration.
Time Frame: From registration to 5 years
Population: Eligible and started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 92
percentage of participants | 92.2 [86.7 to 97.8]

4. Secondary Outcome: Percentage of Participants Alive Without Disease (Disease-free Survival)
Description: An event for disease-free survival is defined as local progression, distant progression, biochemical failure, initiation of salvage hormone therapy, or death due to any cause.Biochemical failure is defined as a rise in prostate-specific antigen (PSA) by at least 2 ng/mL over the current nadir. Local progression is defined as documented progressive disease on digital rectal examination or a post-implant prostate biopsy showing carcinoma. Distant progression is defined as documented lymphatic or hematogenous metastatic disease. Disease-free survival time is defined as time from registration to the date of first event or last known follow-up (censored). Disease-free survival rates are estimated using the Kaplan-Meier method. Analysis occurred after all participants were potentially observed for at least 5 years from registration.
Time Frame: From registration to 5 years
Population: Eligible and started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 92
percentage of participants | 61.2 [51.1 to 71.3]

5. Secondary Outcome: Percentage of Participants With Prostate Cancer Death at 5 Years (Disease-specific Survival)
Description: An event for prostate cancer death is defined as any of the following: primary cause of death certified as due to prostate cancer, death associated with tumor progression occurring after initiation of salvage anti-tumor therapy, death associated with a rise in the serum PSA level on at least two consecutive occasions that occurs during or after salvage androgen suppression therapy, death associated with disease progression in the absence of any anti-tumor therapy, or death from a complication of protocol therapy irrespective of disease status. Time to prostate cancer death is defined as time from registration to date of first event, last known follow-up (censored), or death unrelated to prostate cancer (competing risk). Prostate cancer death rates are estimated using the cumulative incidence method. Analysis occurred after all participants were potentially observed for at least 5 years from registration.
Time Frame: From registration to 5 years
Population: Eligible and started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 92
percentage of participants | 92.2 [86.7 to 97.8]

6. Secondary Outcome: Percentage of Participants With Local Failure at 5 Years
Description: Local progression is defined as documented progressive disease on digital rectal examination or a post-implant prostate biopsy showing carcinoma. Time to local failure is defined as time from randomization to the date of first local failure, last known follow-up (censored), or death without local failure (competing risk). Local failure rates are estimated using the cumulative incidence method. Analysis occurred after all patients were potentially observed for at least 5 years from registration.
Time Frame: From registration to 5 years
Population: Eligible and started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 92
percentage of participants | 3.3 [0.9 to 8.6]

7. Secondary Outcome: Percentage of Participants With Distant Failure at 5 Years
Description: Distant failure is defined as documented lymphatic or hematogenous metastatic disease. Time to distant failure is defined as time from registration to the date of first distant failure, last known follow-up (censored), or death without distant failure (competing risk). Distant failure rates are estimated using the cumulative incidence method. Analysis occurred after all participants were potentially observed for at least 5 years from registration.
Time Frame: From registration to 5 years
Population: Eligible and started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 92
percentage of participants | 10.0 [4.9 to 17.2]

8. Secondary Outcome: Percentage of Participants With Biochemical Failure at 4 Years
Description: Biochemical failure is defined as PSA 2 ng/ml or more higher than the nadir PSA value, or initiation of hormone therapy at any time after brachytherapy. (If the PSA rise is within 36 months following brachytherapy and is followed by a subsequent non-hormonal induced PSA decrease, the patient will not be considered as a failure.) Time to biochemical failure is defined as time from registration to the date of first biochemical failure, last known follow-up (censored), or death without local recurrence (competing risk). Biochemical failure rates are estimated using the cumulative incidence method. Analysis occurred after all participants were potentially observed for at least 5 years from registration.
Time Frame: From registration to 5 years
Population: Eligible and started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brachytherapy
Number analyzed (Participants) | 92
percentage of participants | 32.2 [22.8 to 42.0]

ADVERSE EVENTS:
Time Frame: 1, 3, 6, 9, and 12 months following implant, then every 6 months for years 2-5, then annually. Maximum follow-up at time of analysis was 11.2 years.
Arm/Group | Brachytherapy
Serious Adverse Events (participants affected / at risk) | 8/92
Other Adverse Events (participants affected / at risk) | 89/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brachytherapy (N=92)
Diarrhea (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Prostate infection [with unknown ANC] (Infections and infestations) | 1
Cystitis (Renal and urinary disorders) | 1
Hemorrhage urinary tract (Renal and urinary disorders) | 1
Urethral obstruction (Renal and urinary disorders) | 1
Urethral stricture (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urogenital disorder (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brachytherapy (N=92)
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 15
Fecal incontinence (Gastrointestinal disorders) | 10
Proctitis (Gastrointestinal disorders) | 15
Rectal hemorrhage (Gastrointestinal disorders) | 23
Rectal pain (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 29
Urinary tract infection [with unknown ANC] (Infections and infestations) | 7
Libido decreased (Psychiatric disorders) | 23
Bladder hemorrhage (Renal and urinary disorders) | 8
Bladder pain (Renal and urinary disorders) | 21
Bladder spasm (Renal and urinary disorders) | 9
Cystitis (Renal and urinary disorders) | 33
Hemorrhage urinary tract (Renal and urinary disorders) | 23
Urethral hemorrhage (Renal and urinary disorders) | 7
Urethral obstruction (Renal and urinary disorders) | 9
Urethral pain (Renal and urinary disorders) | 15
Urethral stricture (Renal and urinary disorders) | 7
Urinary frequency (Renal and urinary disorders) | 83
Urinary incontinence (Renal and urinary disorders) | 58
Urinary retention (Renal and urinary disorders) | 55
Urogenital disorder (Renal and urinary disorders) | 17
Ejaculation disorder (Reproductive system and breast disorders) | 15
Erectile dysfunction (Reproductive system and breast disorders) | 54
Prostatic pain (Reproductive system and breast disorders) | 6
Hot flashes (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.